CLINICAL TRIAL: NCT07033455
Title: A Phase 1, Open-label Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of HRS-1893 in Healthy Participants
Brief Title: A Trial of HRS-1893 in Healthy Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HRS-1893-105
Record Dates: First submitted 2025-05-20; First posted 2025-06-24 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-06

CONDITIONS: Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Intervention Model Description: HRS-1893 Oral dosage only
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-1893 Dose level 1 (Experimental): Single oral low dose of HRS-1893 (dose level 1)
  Interventions: Drug: HRS-1893
- HRS-1893 Dose level 2 (Experimental): Single oral high dose of HRS-1893 (dose level 2)
  Interventions: Drug: HRS-1893

INTERVENTIONS:
Drug: HRS-1893 — Single dose of HRS-1893 orally administered

SUMMARY:
The purpose of this study is to assess the safety and PK characteristics of a single oral dose of HRS-1893 in healthy voluunters.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy white participants;
2. Ability to understand the trial procedures and possible adverse events, volunteer to participate in the trial, and provide written informed consent, be able to comply with all the requirements, and able to complete the study.
3. Male aged between 18 to 55 years of age (inclusive)
4. Women with body weight ≥ 45.0 kg, men with body weight ≥ 50.0 kg, body mass index (BMI) between 19.0 and 30.0 kg/m2 (inclusive) at screening.
5. Negative pregnancy test for women of childbearing potential (WOCBP) at baseline. Men and WOCBP must agree to take highly effective contraceptive methods

Exclusion Criteria:

1. History or evidence of clinically significant disorders
2. History of cardiomyopathy and/or unexplained heart failure
3. Individuals with a history of drug allergies, specific allergies
4. Any other circumstances (e.g., not suitable for venous access) or laboratory abnormality that, in the investigator's judgment, may increase the risk to the participant, or be associated with the participant's participation in and completion of the study or could preclude the evaluation of the participant's response.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2025-06-25 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
PK profile of HRS-1893 after a single oral (PO) administration | Day 8
  Pharmacokinetics PK Cmax: Plasma Cmax
PK profile of HRS-1893 after a single oral (PO) administration | Day 8
  Pharmacokinetics PK AUClast : Plasma AUClast
PK profile of HRS-1893 after a single oral (PO) administration | Day 8
  Pharmacokinetics PK AUC0-inf: Plasma AUC0-inf
PK profile of HRS-1893 after a single oral (PO) administration | Day 8
  Pharmacokinetics PK Tmax :Plasma Tmax
PK profile of HRS-1893 after a single oral (PO) administration | Day 8
  Pharmacokinetics PK t1/2 : Plasma t1/2
PK profile of HRS-1893 after a single oral (PO) administration | Day 8
  Pharmacokinetics PK CL/F: Plasma CL/F
PK profile of HRS-1893 after a single oral (PO) administration | Day 8
  Pharmacokinetics PK Vz/F: Plasma Vz/F
Cumulative amount of drug excreted in urine of HRS-1893 after a single oral administration | Day 8
  Cumulative amount of drug excreted in urine (Ae,ur)
Cumulative percentage of dose recovered in urine of HRS-1893 after a single oral administration: | Day 8
  Cumulative percentage of dose recovered in urine (%Ae,ur)
Renal clearance of HRS-1893 after a single oral administration | Day 8
  Renal clearance (CLr)

SECONDARY OUTCOMES:
Safety and Tolerability Based on Incidence and Severity of Treatment Emergent Adverse Events | Day 8
  Number of participants with Adverse events and Serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Linear Clinical Research, Nedlands, Western Australia, Australia